CLINICAL TRIAL: NCT00070941
Title: SAM-e Treatment of Depression in Parkinson's Disease.
Brief Title: SAM-e for the Treatment of Depression in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: R01AT000941-01A1 (NIH); R01AT000941-01A1 (NIH); 075255364 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2003-10-09; First posted 2003-10-13 (Estimated); Results first posted 2016-07-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-06

CONDITIONS: Parkinson's Disease; Depression
Keywords: Parkinsons Disease; Depression; SAM-e
MeSH Terms: conditions — Parkinson Disease; Depression | interventions — S-Adenosylmethionine; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SAM-e (Experimental): 40 subjects receiving oral SAM-e, 1200mg or 1800mg daily in two divided doses, and placebo escitalopram.
  Interventions: Drug: SAM-e
- Escitalopram (Active Comparator): 40 subjects receiving oral escitalopram 20mg or 40 mg daily, in two divided doses, and placebo SAM-e.
  Interventions: Drug: oral escitalopram
- Placebo Comparator (Placebo Comparator): 20 subjects receiving oral placebo escitalopram and placebo SAM-3 daily in two divided doses.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SAM-e — oral SAM-e in two divided doses, 1200mg or 1800mg daily, with placebo escitalopram.
  Other Names: 1 Experimental
  Arms: SAM-e
Drug: oral escitalopram — 20mg or 30mg daily in two divided doses, along with placebo SAM-e.
  Arms: Escitalopram
Drug: placebo — oral placebo escitalopram and oral placebo SAM-e daily in two divided doses.
  Arms: Placebo Comparator

SUMMARY:
This study will test a chemical called s-adenosyl-methionine (SAM-e) for the treatment of depression in patients with Parkinson's disease (PD).

DETAILED DESCRIPTION:
PD is commonly associated with depression, but conventional antidepressants have limited efficacy in patients with PD and may exacerbate motor symptoms. SAM-e is available in the United States as a food supplement and is promoted as a mood enhancer. SAM-e improves dopamine transmission, may have a beneficial effect on dopamine receptors, and may be a good alternative to the currently-used antidepressants in patients with PD. This study will investigate whether SAM-e is safe and effective in the treatment of depression associated with PD. The efficacy of SAM-e will be compared to placebo and to escitalopram, a selective serotonin reuptake inhibitor commonly used for the treatment of depression in PD.

Participants in this study will be randomly assigned to receive SAM-e, escitalopram, or placebo for 12 weeks. Some participants may choose to extend treatment for an additional 12 weeks (for a total of 24 weeks on study medication). Participants will have study visits at entry and Weeks 2, 4, 8, and 12. Study visits will include neurological evaluation, psychiatric evaluation, blood tests, and quality of life questionnaires. A telephone interview will be conducted at Week 10.

ELIGIBILITY:
Inclusion Criteria

* Idiopathic Parkinson's disease as indicated by the presence of at least two of the following signs: resting tremor, rigidity, bradykinesia, or postural reflex impairment
* Stable anti-parkinson medication regimen, with no change in medications in the 4 weeks prior to study entry
* No antidepressant or antipsychotic medications within 30 days prior to study entry
* Agree not to start other pharmacotherapy, psychotherapy, or behavior therapy while participating in the trial
* Acceptable methods of contraception
* Ability to read and/or follow written and oral instructions presented in English
* Sufficient cognitive ability (baseline Mini-Mental Status > 24) to provide informed consent

Exclusion Criteria

* History of cardiac, hepatic, renal, hematologic, respiratory, endocrine, vascular, metabolic, or other systems abnormalities that are clinically relevant in the opinion of study officials
* Certain abnormal laboratory values
* Pregnant or breastfeeding
* Use of an investigational drug within 3 months of study entry
* Use of St. John's Wort or any other "natural" product known to have mood enhancing properties in the 30 days prior to study entry
* Selegiline or other monoamine oxidase inhibitor within the 6 weeks prior to study entry
* Regular usage of anti-anxiety medications or habitual use of sleep medications, although occasional use of certain hypnotics (temazepam, melatonin, or zolpidem) is allowed
* Psychotherapy initiated in the 6 months prior to study entry
* History of bipolar disorder, hypomania, mania, schizophrenia, or other psychotic disorder
* Serious suicidal attempt in the 12 months prior to study entry or serious suicidal tendencies/potential
* Use of dopamine receptor antagonist (metoclopramide, haloperidol)
* Secondary Parkinsonian symptoms due to drugs (including dopamine receptor antagonists), metabolic disorders, cerebrovascular disease, encephalitis, or other degenerative diseases

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2003-07; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Di Rocco, MD, Principal Investigator — NYU
Locations (1):
- New York University, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment dates 01NOV2006-31OCT2008 locations: James Godbold, PH.D. Mount Sinai School of Medicine Steven Ferrando, MD - Weill Medical College of Cornell University Teodoro Bottiglieri, Ph.D. - Baylor College of Medicine Dr. Peter Werner - Albert Einstein College of Medicine
Groups:
- SAM-e: SAM-e, 1200mg or 2400 mg
- Escitalopram: oral Escitalopram 10mg or 20m
- Placebo Comparator: oral placebo Escitalopram and placebo SAM-e
Period: Overall Study
Arm/Group | SAM-e | Escitalopram | Placebo Comparator
Started | 12 | 11 | 6
Completed | 2 | 3 | 2
Not Completed | 10 | 8 | 4
Not completed — Adverse Event | 10 | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- SAM-e: oral SAM-e, 1200mg or 2400 mg
- Total: Total of all reporting groups
Arm/Group | SAM-e | Escitalopram | Placebo Comparator | Total
Number analyzed (Participants) | 12 | 11 | 6 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 0 | 9
  >=65 years | 6 | 8 | 6 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 3 | 14
  Male | 6 | 6 | 3 | 15
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 6 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Depression Scale
Description: very severe, >23/29; severe, 19-22/29; moderate, 14-18/29; mild, 8-13/29; and no depression, 0-7/29 (Hamilton M., J Neurol Neurosurg Psychiatry. 1960 Feb;23:56-62.)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SAM-e | Escitalopram | Placebo Comparator
Number analyzed (Participants) | 12 | 8 | 4
units on a scale
  Baseline Visit Measurement | 17 (4.8) | 17.5 (5.4) | 20.7 (3.2)
  Week 12 Measurement | 11.4 (7.3) | 5.3 (3.3) | 16.2 (3.6)

ADVERSE EVENTS:
Groups:
- SAM-e: Group A/Forty patients receiving oral SAM-e, 1200mg or 2400 mg
- Oral Escitalopram: Group B/Forty patients receiving oral Escitalopram 10mg or 20m
- Placebo: Group C/Twenty patients receiving oral placebo Escitalopram an
Arm/Group | SAM-e | Oral Escitalopram | Placebo
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/11 | 3/6
Other Adverse Events (participants affected / at risk) | 12/12 | 8/11 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SAM-e (N=12) | Oral Escitalopram (N=11) | Placebo (N=6)
Hypotension Orthostatic (Vascular disorders) | 1 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SAM-e (N=12) | Oral Escitalopram (N=11) | Placebo (N=6)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 0 | 0
AGITATION (Psychiatric disorders) | 3 | 1 | 1
ANOREXIA (Metabolism and nutrition disorders) | 5 | 2 | 2
ANXIETY (Psychiatric disorders) | 1 | 0 | 0
APPETITE DECREASED (Metabolism and nutrition disorders) | 0 | 1 | 0
BALANCE DIFFICULTY (Ear and labyrinth disorders) | 0 | 2 | 0
BLOATING (Gastrointestinal disorders) | 0 | 1 | 0
BLOOD PRESSURE INCREASED (Vascular disorders) | 0 | 0 | 1
CHEST PAIN (Cardiac disorders) | 1 | 0 | 0
CONFUSION (Psychiatric disorders) | 2 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 6 | 2 | 3
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 0 | 1
DIZZINESS (Nervous system disorders) | 2 | 4 | 3
DROWSINESS (Nervous system disorders) | 4 | 2 | 2
DYSKINESIA (Nervous system disorders) | 0 | 0 | 1
EXCITABILITY (Psychiatric disorders) | 1 | 0 | 1
FAINTNESS (Nervous system disorders) | 1 | 3 | 3
FALL (Injury, poisoning and procedural complications) | 2 | 1 | 2
HALLUCINATION AUDITORY (Psychiatric disorders) | 0 | 0 | 1
HALLUCINATION VISUAL (Psychiatric disorders) | 0 | 0 | 2
HEADACHE (Nervous system disorders) | 3 | 4 | 1
HYPOTENSION ORTHOSTATIC (Vascular disorders) | 1 | 0 | 1
INDIGESTION (Eye disorders) | 0 | 1 | 0
INSOMNIA (Psychiatric disorders) | 4 | 3 | 5
LEG PAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0
LETHARGY (Nervous system disorders) | 1 | 0 | 0
LIBIDO DECREASED (Psychiatric disorders) | 1 | 0 | 0
MOUTH DRY (Gastrointestinal disorders) | 3 | 4 | 3
MUSCLE RIGIDITY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 4 | 3 | 5
PAIN (General disorders) | 0 | 1 | 0
POLYCYTHAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 1
STOMACH UPSET (Gastrointestinal disorders) | 1 | 0 | 0
SYNCOPE (Nervous system disorders) | 1 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 2 | 1
TREMOR (Nervous system disorders) | 4 | 3 | 2
TREMOR COARSE (Nervous system disorders) | 0 | 0 | 1
URINARY FREQUENCY (Renal and urinary disorders) | 1 | 0 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 0 | 1
VISION BLURRED (Eye disorders) | 2 | 5 | 2
VIVID DREAMING (Psychiatric disorders) | 1 | 0 | 0
VOMITING (Gastrointestinal disorders) | 1 | 0 | 1
WEAKNESS GENERALIZED (General disorders) | 2 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
According to the NIH -grant that supported this clinical trial all publications must be reported to the grant office prior to the release of publications.

Statement from NIH award letter:

This includes manuscripts submitted or accepted for publication to the awarding component. Report only those publications resulting directly from this grant and those publications. If there have been no publications, so state.